CLINICAL TRIAL: NCT00302783
Title: Randomized Controlled Trial of Multi-Source Feedback to Pediatric Residents: The Formative Value of an ACGME Competency-Based Assessment Tool.
Brief Title: Randomized Controlled Trial of Multi-Source Feedback to Pediatric Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Ambulatory Pediatric Association (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: 03-12-37X
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2006-03-15 (Estimated); Status verified 2006-01

CONDITIONS: Education, Medical; Education, Competency-Based; Feedback; Communication; Humanism
Keywords: Education, Medical; Education, Competency-Based; Multi-Source Feedback; Communication; Professionalism
MeSH Terms: conditions — Communication

INTERVENTIONS:
Behavioral: Multi-Source Feedback: including self-assessment & coaching

SUMMARY:
The purpose of this study is to test whether multi-source feedback, including self-assessment and tailored coaching, improves resident communication skills and professionalism. We hypothesize that residents who are assigned to receive multi-source feedback, in addition to receiving standard feedback, will improve significantly more than residents receiving standard feedback alone, as measured by parent and nurse ratings of specific behaviors over time.

ELIGIBILITY:
Inclusion Criteria:

* Residents entering their first year of training
* Scheduled for the two pediatric inpatient rotations where parent and nurse evaluations would be collected

Exclusion Criteria:

* Residents from combined Internal Medicine/Pediatric training programs

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 2004-06; Study Completion 2005-09

PRIMARY OUTCOMES:
The difference between groups in the change in parent and nurse ratings of specific communication skills and professionalism behaviors from baseline to follow-up (average 5 months later)

CONTACTS AND LOCATIONS:
Overall Officials: William B Brinkman, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Brinkman WB, Geraghty SR, Lanphear BP, Khoury JC, Gonzalez del Rey JA, Dewitt TG, Britto MT. Effect of multisource feedback on resident communication skills and professionalism: a randomized controlled trial. Arch Pediatr Adolesc Med. 2007 Jan;161(1):44-9. doi: 10.1001/archpedi.161.1.44. PMID 17199066